CLINICAL TRIAL: NCT06688500
Title: Bowel Dysfunction and HoLEP Outcomes
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Krambeck, Urologic Surgeon, Northwestern University
Other Study IDs: STU00220105
Record Dates: First submitted 2024-06-26; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Urologic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bowel function post Holmium Laser Enucleation of the Prostate — Observing post operative bowel functions among participants who have undergone a HoLEP procedure.

SUMMARY:
The objective of this prospective study is to examine the correlation and effects of bowel dysfunction on outcomes for patients undergoing holmium laser enucleation of prostate (HoLEP) for lower urinary tract symptoms secondary to benign prostatic hyperplasia (BPH).The investigator hypothesizes that patients who have more bowel dysfunction based on higher severity scores on patient-reported validated questionnaires will experience more symptoms in the immediate post-operative period and may have slower recovery of urinary control. Assessment of pre, peri, and post-procedural bowel dysfunction via the Constipation Severity Score (CSS) and Vaizey Incontinence Questionnaire will aid the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Males18-89 undergoing HoLEP
* Able to read, understand, and complete patient questionnaires
* Willing to sign the informed consent form

Exclusion Criteria:

* Patients with bowel diversion (colostomy, ileostomy)
* Patients with known neurogenic bowel
* Patients having concurrent ureteroscopy+/-laser lithotripsy, percutaneous nephrolithotomy, or non-urologic surgery at time of HoLEP
* Anticipated need for perineal urethrostomy at time of HoLEP
* Prior pelvic radiation or patients with history of bladder cancer with or without Bacillus Calmette-Guerin (BCG) therapy
* Patients who lack decisional capacity

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients 18-89 years old undergoing HoLEP
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Difference in American Urologic Association Symptom Score (AUASS) | 3 months
  Identifying differences in AUASS scores pre-operatively versus post-operatively. An AUA symptom score of 0-7 is considered mild, 8-19 is moderate, and 20-35 is severe. This will be used in combination with the other measures to come up with total severity of overall condition.
Collecting preoperative bowel dysfunction scores via Constipation Severity Scale (CSS) and Vaizey Incontinence questionnaires | 3 months
  Identifying differences in CSS/Vaizey Incontinence questionnaires at pre-op 3- month clinic follow-up. Minimum score of 0 indicates perfect continence versus 24 which indicates total incontinence. This will be used in combination with the other measures to come up with total severity of overall condition.

SECONDARY OUTCOMES:
Change between pre-operative and post-operative bowel dysfunction scores and symptoms | 6 months
  Identifying changes in symptom management/resolve: post-op retention, time with catheter, gross hematuria, Urinary Tract Infection, Emergency Department visits and any other complications. This will be used in combination with the other measures to come up with total severity of overall condition.
Monitoring efficacy of procedure | 1 year
  Identifying changes with post void residual, Michigan Incontinence Score Index (MISI). With a score range of 0-32, identifying severity and total bother. This will be used in combination with the other measures to come up with total severity of overall condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No